CLINICAL TRIAL: NCT01320267
Title: Single Incision Laparoscopic Right Hemi-colectomy Pilot Study
Brief Title: Single Port Laparoscopic Colectomy
Acronym: SILS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Industry Funding Withdrawn
Sponsor: University of British Columbia (Other)
Collaborators: Tyco Healthcare Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H10-00969
Record Dates: First submitted 2011-03-01; First posted 2011-03-22 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Colon Cancer
Keywords: Resectable right colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SILS right hemicolectomy (Experimental): Single arm with intervention only.
  Interventions: Procedure: Single port laparoscopic right hemicolectomy

INTERVENTIONS:
Procedure: Single port laparoscopic right hemicolectomy — above procedure using Roticulating instruments (from Covidien)

SUMMARY:
The investigators will document the success for completing laparoscopic resection of cancer in the right colon using a new single port access technique. The current procedure requires 4 incisions for 4 separate ports. With technological advancement of newly designed instruments it is now possible to do the same laparoscopic procedure through a single port. The investigators want to demonstrate here in British Columbia that it is a safe procedure with similar success and outcomes compared to the standard 4-port laparoscopic operation.

The investigators propose that this procedure may provide early discharge due to less pain and also be associated with less wound infection and hernia complications. The single incision will have improved cosmesis compared to the standard 4-port standard laparoscopic procedure.

DETAILED DESCRIPTION:
Purpose:

The purpose of the study is to demonstrate that single port right hemi-colectomy can be performed with consistency. The second purpose is to assess single port surgery in terms of length of stay in the hospital, analgesics requirement, and length of scar at 30 days. The single port surgery is a latest advancement towards achieving minimal scarring after major abdominal surgery.

Justification:

Laparoscopic Colon resection is well-documented and standard practice in many centers throughout the world. A Cochrane Review of 25 Randomized Control Trials (RCT) published in 2005 looked at the short term (30 Days) benefits of laparoscopic colorectal resection showed better outcome in intra-operative blood loss, intensity of postoperative pain, postoperative hospital stay, duration of postoperative ileus, and pulmonary functions (1). Total morbidity and local (surgical) morbidity was decreased in the laparoscopic groups. Until the 30th postoperative day, quality of life was better in laparoscopic patients. They concluded if the long-term oncological results of laparoscopic and conventional resection of colonic carcinoma show equivalent results, the laparoscopic approach should be preferred in patients suitable for this approach to colectomy. A Cochrane Review published in 2008 looked at 33 RCT's comparing laparoscopic/Laparoscopic-assisted and open colectomy for colo-rectal carcinoma found similar long-term oncologic outcomes in both groups (2).

Single Incision Laparoscopic Surgery (SILS) instead of traditional 4 ports theoretically may reduce the wound complications. For cholecystectomy, a blinded randomized control study showed significant reduction in pain control at sub-costal port-sites in 2-port versus 4-port laparoscopic cholecystectomy and also showed similar pain at umbilical port (3).

There have been few reports of performing colectomy through a single port similar to the SILS cholecystectomy as mentioned above. Remzi et al published a report of performing sigmoid-colectomy for polyp using single umbilical tri-port system (4). Merchant et al used a single port (this time a Gel-port) to perform SILS right hemicolectomy (5). Bucher reported a case of single incision laparoscopic sigmoidectomy for stenosis due to endometriosis (6). They questioned if SILS colectomy offers benefits except in cosmesis, when compared to standard laparoscopic surgery.

The above-mentioned publications of SILS colectomy used conventional and not so conventional instruments (curved and/or articulating forceps). The availability of these instruments due to technical advancement has opened the door for these procedures to be performed more routinely. In a recent study this technique was applied effectively and performed in comparable operative times to traditional 3-port cholecystectomy with a learning curve of approximately 5 cases (7).

Recently Dixon et al.(8) demonstrated by performing variety of colo-rectal procedures using a single port laparoscopic technique. They performed, right hemi-colectomy, extended right hemi-colectomy, total colectomy with ileo-anal anastomosis, procto-colectomy, restorative procto-colectomy with ileo-anal pouch formation and anterior resection. Two of these procedures were for cancers. All operations were performed using a single incision tri-port system with harmonics scalpel, linear/circular stapler and standard laparoscopic instruments.

Methods:

The investigators will assess short-term outcome variables for the single incision laparoscopic resection procedure in a pilot study of 20 patients diagnosed with resectable right colon cancer. The investigators will compare these short term outcome variables to an aggregate group of patients that previously had undergone standard 4-port laparoscopic resection of right colon cancer in a 12-month period (2009).

The outcome variables are:

1. Successful completion of the right hemicolectomy
2. Use of additional ports and reason
3. Conversion to an open procedure and reason
4. Duration of the surgery
5. Operative complications
6. Number and total length of surgical incisions
7. Postoperative analgesia requirements
8. Postoperative complications
9. Length of postoperative hospital stay
10. Cancer stage (TNM)
11. Resection margin clearance
12. Number of lymph nodes assessed

Data collection:

Data will be collected prospectively for patients undergoing the single port laparoscopic resection. Data will be abstracted retrospectively from electronic hospital and office charts for patients that previously had standard laparoscopic resection of right colon cancer.

Statistical analysis:

Demographic, operative and postoperative data will be summarized and reported as counts and percents for categorical variables and Mean ± Standard Deviation (plus Median & Min. Max.) for continuous variables. Outcomes of the two groups will be compared by independent samples t-tests and non-parametric median tests for continuous variables and Chi-square or Fisher's exact tests for categorical variables.

Sample size:

The pilot study sample size of 20 was chosen on the basis of a reasonable number of patients to be recruited in one year. The comparison group size for patients previously having standard laparoscopic resection was chosen only for convenience but is estimated at approximately 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 19 years or older diagnosed with resectable right colon cancer

Exclusion Criteria:

* Advanced cancer on routine preoperative CT (local invasion, distant metastases)
* maximum diameter of cancer > 5cm
* previous abdominal surgery
* emergency surgery
* pregnancy
* ages < 18 years old
* ASA (American Society of Anesthesiologists) Class III or above
* Any other contraindications to laparoscopic surgery
* Non-English speaking/reading or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Successful completion of the right hemicolectomy | 1 day
  The first and main outcome is to assess if right hemicolectomy can be safely performed using the Single Port.

SECONDARY OUTCOMES:
Use of additional ports and reason | 1 day
  This is to see that even using roticulating laparoscopic instruments, how often and how many additional ports were placed.
Conversion to an open procedure and reason | 1 day
Duration of surgery | 1 Day
Operative complications | 1 Day
  this includes, bleeding complications and inadvertant bowel or other abdominal visceral injury.
Total Length of surgical incision (cm) | 30 days
Postoperative analgesia requirements (total opioid used) | 30 days
  total mg of Morphine used. If morphine is not used and alternative opioid used, this will be coverted standard conversion to equivalent dose of Morphine.
30 Day Mortality | 30 Days
Length of postoperative hospital stay | 30days
Pathological Cancer stage (TNM) | 15 Days
Pathology: Resection margin clearance | 15 Days
Number of lymph nodes assessed | 15 Days
Total Number of Surgical Incisions | 1 Day
Wound Infection | 30 Days
  yes/no, Deep Surgical site infection vs Superficial Surgical site infection.
Postoperative complications: Requirement of Re-operation | 30 Days
  Yes/NO
Postoperative complications: Reason for reoperation | 30 Days
  (if needed re-operation)
Postop Complications: Wound Dehiscence | 30 Day
Postoperative Complications: Others | 30 Day
  including deep vein thrombosis/pulmonary embolism (DVT/PE), myocardial infarction, stroke and pneumonia
30 Day Re-admission | 30 Days
Postoperative Measure of Pain | 3 DAYS
  Visual Analogue Scale to quantify pain on POD#1, #2 AND #3